CLINICAL TRIAL: NCT05215275
Title: Comparison of Different Exercise Trainings on Heart Rate Variability in Community Residents With Higher Visceral Adipose Tissue
Brief Title: Comparison of Different Exercise Trainings on Heart Rate Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Tainan Junior College of Nursing (Other)
Responsible Party: Principal Investigator, Yu-Hsuan Chang, assistant professor, National Tainan Junior College of Nursing
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 109-516
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Fat Burn; Exercise
Keywords: heart rate variability; visceral adipose tissue; exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MICT to HIIT (Experimental): participants will receive moderate-intensity continuous training lasting 8 weeks, and then exchange to high-intensity interval training lasting 8 weeks, with 8 weeks rest insert to two different modalities of exercise.
  Interventions: Behavioral: exercise
- HIIT to MICT (Experimental): participants will receive high-intensity interval training lasting 8 weeks, and then exchange to moderate-intensity continuous training lasting 8 weeks, with 8 weeks rest insert to two different modalities of exercise.
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — the exercise consists of two different modalities: moderate-intensity continuous training (MICT): the main MICT program will be designed to last 30 minutes. The MICT will be designed to involve core muscle training (e.g., march, step touch, lunge, V-step, box step, twist, knee up, scoop, and scissors).
  high-intensity interval training (HIIT): The HIIT motions will be a mix of spiderman mountain climbers, standing oblique crunches, squats, froggers, jumping jacks, foot fire, jump squats, and mountain climbers. A total of four sets will be performed with 1-minute rests between sets. Each set comprises eight motions, with each motion lasting 30 seconds and a rest interval of 10 seconds between motions. Participants in the HIIT group will perform the most repetitions possible within 30 seconds.

SUMMARY:
The aims of this project are to compare the effects between 8-week moderate-intensity continuous training (MICT) and high-intensity interval training (HIIT) on improving HRV.

DETAILED DESCRIPTION:
Background: Both heart rate variability (HRV) and visceral adipose tissue (VAT) are crucial factors predicting cardiovascular diseases, and both can be improved by exercise training. HRV can provide information regarding sympathetic and parasympathetic activity. Studies have demonstrated that HRV and VAT are correlated. VAT accumulation may dysregulate the balance of the sympathetic and parasympathetic nervous system. However, the correlation between sympathetic activation and VAT is controversial and limited by a paucity of studies, and the optimal exercise modality for improving HRV remains debatable. Therefore, the aims of this 1-year project are to compare the effects between 8-week moderate-intensity continuous training (MICT) and high-intensity interval training (HIIT) on improving HRV.

Methods: Purposive sampling will be used to enroll at least 72 community residents aged 40-64 years with VAT over 100 cm2. A two-phase crossover design will be used to understand the change patterns of HRV and VAT in the 8-week different exercise phase and with 8-week washout period insertion. Participants will initially be randomized into either the MICT or HIIT group for 8 weeks, and the groups will then be exchanged for the later 8 weeks. HRV parameters and VAT will be measured at four time points at baseline (T0), the end of the first phase (8-week later, T1), the initial of second phase (16-week later, T2), and the end of the second phase (24-week later, T2). Linear mixed models (LMMs) with random effects will be used to compare the effects of 8-week different exercise modalities on HRV and explore the effect of VAT changes on HRV over the 24-week intervention.

Relevance to clinical practice: The results of this study can reveal the optimal exercise modality for improving HRV among community residents with higher VAT and clarify HRV and VAT change patterns in exercise and rest phase and the correlation between HRV and VAT. These findings would provide evidence that clinical health professionals can use to promote health benefits through exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Community residents (a) who are 40-64 years old, (b) with a VAT of ≧ 100 cm2 measured using a body composition analyzer, and (c) who can communicate in Mandarin or Taiwanese will be included.

Exclusion Criteria:

* This study will exclude (a) residents with recent unstable conditions (stroke, cardiovascular and respiratory diseases, handicap, pregnancy, mental disorders, systolic blood pressure > 200 mmHg, or diastolic blood pressure > 110 mmHg), (b) residents with contraindications to body composition analyzer measurement (e.g., people with pacemakers, artificial metal joints, and amputated hands or feet) and residents who cannot stand during testing, and (c) residents with habits or lifestyles that may affect HRV (e.g., smoking or alcohol abuse and shift work).

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
visceral adipose tissue | four times (baseline, 8-week, 16-week, 24-week)
  explore which modality of exercise can reduce the greatest area of visceral adipose tissue under body compostion analyzer measurement

SECONDARY OUTCOMES:
heart rate variability | four times (baseline, 8-week, 16-week, 24-week)
  explore the trajectory of heart rate variability among two groups of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsuan Chang, phD, Principal Investigator — National Tainan Junior College of Nursing
Locations (1):
- National Tainan Junior College of Nursing, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No